CLINICAL TRIAL: NCT05866185
Title: Improving Adherence to Evidence-Based Practice Using an Innovative and Easy-to-Use Health IT Solution
Brief Title: Improving Adherence to Homework During Therapy
Acronym: Adherely STTR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 002555; 5R41MH126734-02 (NIH)
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Results first posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Anxiety; Depression; Depression/Anxiety
Keywords: mhealth; mental health; adult mental health; homework; health technology
MeSH Terms: conditions — Anxiety Disorders; Depression; Psychological Well-Being | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapy (Active Comparator): Standard regular therapy.
  Interventions: Behavioral: Therapy
- Therapy + Adhere.ly (Experimental): Standard regular therapy, enhanced with Adhere.ly
  Interventions: Behavioral: Therapy + Adhere.ly

INTERVENTIONS:
Behavioral: Therapy — The standard of care procedures for adults with clinically elevated anxiety and/or depression from their mental health provider.
  Arms: Therapy
Behavioral: Therapy + Adhere.ly — Participants receive therapy as usual enhanced with a simple, HIPAA-compliant, web-based application to help mental health providers implement homework during therapy for adults with elevated anxiety and/or depression. The three major components of the app help providers to (1) Practice interactive, digitized therapeutic exercises with patients in-session; (2) Remind patients to practice exercises for homework, and (3) Review homework during the next session.
  Arms: Therapy + Adhere.ly

SUMMARY:
The purpose of this study is to expand Adhere.ly- a simple, HIPAA-compliant, web-based platform to help therapists engage clients in practicing therapeutic skills between sessions (homework) during mental health treatment by conducting a trial comparing standard therapy to therapy enhanced with Adhere.ly.

ELIGIBILITY:
Inclusion Criteria:

Providers:

* English-speaking
* Mental health providers who have obtained at least a master's degree in social work, counseling, clinical psychology, or related field
* Carry active mental health treatment caseloads in the U.S.
* Have a laptop, tablet, or smartphone with internet access

Clients:

* English-speaking
* Treatment-seeking adults ≥18 years
* Clinically elevated anxiety and depression as indicated by a score ≥10 on the GAD-7 and/or PHQ-8
* Have a laptop, tablet, or smartphone with internet access

Exclusion Criteria:

Client with self-reported:

* Active psychotic symptoms (e.g., hallucinations, delusions)
* Significant cognitive disability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian E Bunnell, PhD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: While 40 therapists were enrolled in the trial, they were not assigned to a treatment arm until after their first referred client enrolled in the study. Not all therapists referred clients who enrolled in the study. As a result, the number of therapists allocated to a treatment arm differs from the number enrolled in the study.
Groups:
- Clients - Therapy: Clients assigned to receive standard regular therapy.
  Therapy: The standard of care procedures for adults with clinically elevated anxiety and/or depression from their mental health provider.
- Clients - Therapy + Adhere.ly: Clients assigned to receive standard regular therapy enhanced with Adhere.ly
  Therapy + Adhere.ly: Participants receive therapy as usual enhanced with a simple, HIPAA-compliant, web-based application to help mental health providers implement homework during therapy for adults with elevated anxiety and/or depression. The three major components of the app help providers to (1) Practice interactive, digitized therapeutic exercises with patients in-session; (2) Remind patients to practice exercises for homework, and (3) Review homework during the next session.
- Therapists - Therapy: Therapists assigned to provide standard regular therapy to clients.
  Therapy: The standard of care procedures for adults with clinically elevated anxiety and/or depression from their mental health provider.
- Therapists - Therapy + Adhere.ly: Therapists assigned to provide standard regular therapy enhanced with Adhere.ly to clients.
  Therapy + Adhere.ly: Participants receive therapy as usual enhanced with a simple, HIPAA-compliant, web-based application to help mental health providers implement homework during therapy for adults with elevated anxiety and/or depression. The three major components of the app help providers to (1) Practice interactive, digitized therapeutic exercises with patients in-session; (2) Remind patients to practice exercises for homework, and (3) Review homework during the next session.
Period: Overall Study
Arm/Group | Clients - Therapy | Clients - Therapy + Adhere.ly | Therapists - Therapy | Therapists - Therapy + Adhere.ly
Started | 14 | 25 | 8 | 10
Completed 3-month Post-baseline | 12 | 21 | 0 | 0
Completed Post-Trial Therapist Assessment | 0 | 0 | 4 | 4
Completed | 12 | 21 | 4 | 4
Not Completed | 2 | 4 | 4 | 6
Not completed — Lost to Follow-up | 2 | 4 | 4 | 6

BASELINE CHARACTERISTICS:
Population: A total of 40 therapists were enrolled in the study. A total of 18 providers referred clients that enrolled in the trial and were subsequently randomized to a treatment condition. Data are reported for those providers who were randomized to a treatment condition.
Groups:
- Total: Total of all reporting groups
Arm/Group | Clients - Therapy | Clients - Therapy + Adhere.ly | Therapists - Therapy | Therapists - Therapy + Adhere.ly | Total
Number analyzed (Participants) | 14 | 25 | 8 | 10 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.21 (7.96) | 26.24 (6.97) | 35.00 (23.50) | 27.40 (22.48) | 30.37 (14.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 20 | 7 | 9 | 49
  Male | 1 | 5 | 1 | 1 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 1 | 0 | 12
  Not Hispanic or Latino | 10 | 18 | 7 | 10 | 45
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 4 | 3 | 2 | 13
  White | 10 | 17 | 3 | 7 | 37
  More than one race | 0 | 4 | 1 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 25 | 8 | 10 | 57

OUTCOME MEASURES:

1. Primary Outcome: Generalized Anxiety Disorder-7 (Gad-7)
Description: The Generalized Anxiety Disorder Scale-7 (GAD-7) assesses the severity of anxiety symptoms in adults. The GAD-7 was completed by clients about themselves. Scores range from 0 to 21 with higher scores indicating worse anxiety symptom severity. A score of 8 or greater is generally considered to indicate clinically significant anxiety symptom severity.
Time Frame: Baseline, 3 Months Post Baseline
Population: The Overall Number of Participants Analyzed refers to the number of participants enrolled and randomized to each arm. The number of participants analyzed in rows differs from this number due to participants being lost to contact and withdrawn from the study. The GAD-7 was completed by clients so data are not presented for therapists.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clients - Therapy | Clients - Therapy + Adhere.ly | Therapists - Therapy | Therapists - Therapy + Adhere.ly
Number analyzed (Participants) | 14 | 25 | 0 | 0
units on a scale
  Baseline | 14.86 (3.70) | 12.88 (4.82) |  |
  3 Months Post Baseline: number analyzed (Participants) | 12 | 21 | 0 | 0
  3 Months Post Baseline | 8.33 (5.23) | 7.62 (4.38) |  |

2. Primary Outcome: Patient Health Questionnaire-8 (PHQ-8)
Description: The Patient Health Questionnaire-8 (PHQ-8) assesses the severity of depression symptoms in adults. The PHQ-8 was completed by clients about themselves. Scores range from 0 to 28 with higher scores indicating worse depression symptom severity. A score of 10 or greater is generally considered to indicate clinically significant depression symptom severity.
Time Frame: Baseline, 3 Months Post Baseline
Population: The Overall Number of Participants Analyzed refers to the number of participants enrolled and randomized to each arm. The number of participants analyzed in rows differs from this number due to participants being lost to contact and withdrawn from the study. The PHQ-8 was completed by clients so data are not presented for therapists.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clients - Therapy | Clients - Therapy + Adhere.ly | Therapists - Therapy | Therapists - Therapy + Adhere.ly
Number analyzed (Participants) | 14 | 25 | 0 | 0
units on a scale
  Baseline | 12.57 (3.98) | 13.80 (5.05) |  |
  3 Months Post Baseline: number analyzed (Participants) | 12 | 21 | 0 | 0
  3 Months Post Baseline | 7.50 (5.55) | 9.19 (6.37) |  |

3. Secondary Outcome: Health-Related Quality of Life (HRQOL-14) - Healthy Mental Health Days Index
Description: The Health-Related Quality of Life (HRQOL-14) - Healthy Mental Health Days Index assesses quality of life in terms of the number of days in the past month that clients' feel that their mental health was "not bad." The HRQOL-14 was completed by clients. Respondents report a number from 0 to 30, and the final score indicates better mental health related quality of life.
Time Frame: Baseline, 3 Months Post Baseline
Population: The Overall Number of Participants Analyzed refers to the number of participants enrolled and randomized to each arm. The number of participants analyzed in rows differs from this number due to participants being lost to contact and withdrawn from the study. The HRQOL-14 was completed by clients so data are not presented for therapists.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clients - Therapy | Clients - Therapy + Adhere.ly | Therapists - Therapy | Therapists - Therapy + Adhere.ly
Number analyzed (Participants) | 14 | 25 | 0 | 0
units on a scale
  Baseline | 9.71 (8.15) | 11.44 (7.61) |  |
  3 Months Post Baseline: number analyzed (Participants) | 12 | 21 | 0 | 0
  3 Months Post Baseline | 15.42 (9.59) | 12.38 (8.95) |  |

4. Secondary Outcome: Homework Rating Scale II (HRS II)
Description: The Homework Rating Scale II (HRS II) assesses levels of homework adherence in cognitive behavior therapy. Total scores range from 0 to 4 with higher scores reflecting better homework adherence. The HRS-II was completed by clients each week and total scores were averaged across weeks between Baseline and 3 Months Post Baseline.
Time Frame: Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 9, Week 10, Week 11, Week 12, Average across weeks reported.
Population: The number of participants reported here differs from the number of participants assigned to arms in the Participant Flow due to some participants not completing the HRS-II and others being lost to contact and withdrawn from the study. The HRS-II was completed by clients so data are not presented for therapists.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clients - Therapy | Clients - Therapy + Adhere.ly | Therapists - Therapy | Therapists - Therapy + Adhere.ly
Number analyzed (Participants) | 11 | 19 | 0 | 0
units on a scale | 2.74 (.78) | 2.92 (.74) |  |

5. Secondary Outcome: Assessment of Core CBT Skills (ACCS) - Cognitive Behavioral Therapy Domain
Description: The Assessment of Core Cognitive Behavioral Therapy (CBT) Skills (ACCS) - Cognitive Behavioral Therapy Domain is an observer rated measure of therapist competence in delivering Cognitive Behavioral Therapy-based interventions. Total scores range from 5 to 20 with higher scores reflecting better competence. The ACCS was used to rate 20% of weekly therapy session audio recordings and total scores were averaged across this 20% of sessions.
Time Frame: as for outcome 4
Population: The ACCS was rated for sessions with client participants as the unit of analysis so data are not presented for therapists. Given that 20% of sessions were randomly selected for ratings data are provided only for clients whose sessions were randomly selected.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clients - Therapy | Clients - Therapy + Adhere.ly | Therapists - Therapy | Therapists - Therapy + Adhere.ly
Number analyzed (Participants) | 5 | 12 | 0 | 0
units on a scale | 15.51 (3.47) | 14.15 (4.88) |  |

6. Secondary Outcome: Attitudes Toward Homework Questionnaire (ATHQ) - Positive Homework Effect Scale
Description: The Attitudes Toward Homework Questionnaire (ATHQ) - Positive Homework Effect Scale assesses therapist perceptions of the positive effects of using homework assignments in psychotherapy. The ATHQ was completed by therapists. Scores range from 1-5 with higher scores indicating therapist perceptions of better positive effects of homework.
Time Frame: Baseline, Post-Trial Therapist Assessment
Population: The ATHQ was completed by therapists so data are not provided for clients.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clients - Therapy | Clients - Therapy + Adhere.ly | Therapists - Therapy | Therapists - Therapy + Adhere.ly
Number analyzed (Participants) | 0 | 0 | 8 | 10
units on a scale
  Baseline |  |  | 4.43 (0.45) | 4.27 (0.43)
  Post-Trial Therapist Assessment: number analyzed (Participants) | 0 | 0 | 4 | 4
  Post-Trial Therapist Assessment |  |  | 4.08 (0.56) | 4.14 (0.53)

7. Secondary Outcome: Working Alliance Inventory - Short Revised (WAI-SR)
Description: The Working Alliance Inventory - Short Revised (WAI-SR) assesses therapeutic alliance, defined as a collaborative relationship between a therapist and client. The WAI-SR was completed by clients about their perceived therapeutic alliance with their therapist. Scores range from 12-60 with higher scores indicating better therapeutic alliance.
Time Frame: 3 Months Post Baseline
Population: The number of participants reported here differs from the number of participants assigned to arms in the Participant Flow due to a partial completion of the 3 Months Post Baseline assessment by one participant. The WAI-SR was completed by clients about their perceived therapeutic alliance with their therapist so data are not provided for therapists.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clients - Therapy | Clients - Therapy + Adhere.ly | Therapists - Therapy | Therapists - Therapy + Adhere.ly
Number analyzed (Participants) | 11 | 21 | 0 | 0
units on a scale | 54.09 (4.01) | 49.91 (9.94) |  |

8. Secondary Outcome: Client Satisfaction Questionnaire - 8 (CSQ-8)
Description: The Client Satisfaction Questionnaire - 8 (CSQ-8) assesses the level of clients' satisfaction with their outpatient mental health services. The CSQ-8 was completed by clients. Scores range from 8-32 with higher scores indicating higher levels of satisfaction.
Time Frame: 3 Months Post Baseline
Population: The number of participants reported here differs from the number of participants assigned to arms in the Participant Flow due to a partial completion of the 3 Months Post Baseline assessment by one participant. The CSQ-8 was completed by clients about their satisfaction with therapy so data are not provided for therapists.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clients - Therapy | Clients - Therapy + Adhere.ly | Therapists - Therapy | Therapists - Therapy + Adhere.ly
Number analyzed (Participants) | 11 | 21 | 0 | 0
units on a scale | 30.55 (2.38) | 28.62 (4.52) |  |

9. Secondary Outcome: Assessment of Core CBT Skills (ACCS) - Homework Domain
Description: The Assessment of Core Cognitive Behavioral Therapy (CBT) Skills (ACCS) - Homework Domain is an observer rated measure of therapist competence in implementing homework during Cognitive Behavioral Therapy-based interventions. Total scores range from 5 to 20 with higher scores reflecting better competence. The ACCS was used to rate 20% of weekly therapy session audio recordings and total scores were averaged across this 20% of sessions.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clients - Therapy | Clients - Therapy + Adhere.ly | Therapists - Therapy | Therapists - Therapy + Adhere.ly
Number analyzed (Participants) | 5 | 12 | 0 | 0
units on a scale | 7.35 (4.17) | 10.91 (3.44) |  |

10. Secondary Outcome: Attitudes Toward Homework Questionnaire (ATHQ) - Negative Session Impact Scale
Description: The Attitudes Toward Homework Questionnaire (ATHQ) - Negative Session Impact Scale assesses therapist perceptions of the negative impacts of using homework assignments in psychotherapy. The ATHQ was completed by therapists. Scores range from 1-5 with higher scores indicating therapist perceptions of worse negative impacts of homework.
Time Frame: Baseline, Post-Trial Therapist Assessment
Population: The ATHQ was completed by therapists so data are not provided for clients.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clients - Therapy | Clients - Therapy + Adhere.ly | Therapists - Therapy | Therapists - Therapy + Adhere.ly
Number analyzed (Participants) | 0 | 0 | 8 | 10
units on a scale
  Baseline |  |  | 2.41 (1.07) | 2.14 (0.47)
  Post-Trial Therapist Assessment: number analyzed (Participants) | 0 | 0 | 4 | 4
  Post-Trial Therapist Assessment |  |  | 1.79 (0.57) | 2.16 (0.65)

ADVERSE EVENTS:
Time Frame: Up to 3 months post baseline
Description: Therapists - Therapy and Therapists - Therapy + Adhere.ly arms were not monitored/assessed for deaths and/or adverse events so data are not reported.
Arm/Group | Clients - Therapy | Clients - Therapy + Adhere.ly | Therapists - Therapy | Therapists - Therapy + Adhere.ly
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/25 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/25 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/14 | 0/25 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-13): https://cdn.clinicaltrials.gov/large-docs/85/NCT05866185/Prot_SAP_001.pdf